CLINICAL TRIAL: NCT04869280
Title: Prucalopride (MOTEGRITY®, RESOTRAN®) Pregnancy Exposure Study: A VAMPSS Post-Marketing Surveillance Study of Prucalopride Safety in Pregnancy
Brief Title: Post-Marketing Study of Prucalopride Safety In Pregnancy
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Collaborators: The Organization of Teratology Information Specialists (Other)
Responsible Party: Sponsor
Other Study IDs: TAK-555-5001; EUPAS40231 (Other: EU PAS Register Number)
Record Dates: First submitted 2021-04-16; First posted 2021-05-03 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Chronic Idiopathic Constipation (CIC)
Keywords: Fetal and infant outcomes; Prucalopride; Pregnancy Registry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort-1: Pregnant Women Exposed to Prucalopride Prior to Enrollment: Pregnant women diagnosed with chronic idiopathic constipation (CIC) or irritable bowel syndrome-constipation (IBS-C) who have been exposed to prucalopride during pregnancy and prior to enrollment will be observed.
  Interventions: Other: No Intervention
- Cohort-2: Pregnant Women Not Exposed to Prucalopride: Pregnant women diagnosed with CIC or IBS-C who have not been exposed to prucalopride will be observed.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
This study collects information on pregnant women with ongoing constipation who took prucalopride and those who did not take prucalopride. The main aim of the study is to learn if any medical problems in pregnant women or their infants might be related to taking prucalopride during pregnancy.

Participants are not required to take prucalopride during the study. The study is non-interventional. Women and their infants are followed during pregnancy and for 1 year after pregnancy to collect information on maternal, pregnancy, and infant outcomes.

During the study, participants will be asked questions during 3 telephone interviews; 2 during pregnancy and 1 just after their expected delivery date. Participants who took or are taking prucalopride will be asked more detailed questions about this during these interviews. All information is collected remotely, and no visits to the study site are required.

Also, all participants will be asked to complete a questionnaire about their baby when their baby is about 1 year old.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1: Prucalopride-Exposed (MOTEGRITY, RESOTRAN) Cohort:

* Pregnant women.
* Exposure to MOTEGRITY or RESOTRAN (generic forms of prucalopride not allowed) for the treatment of chronic idiopathic constipation (CIC) or irritable bowel syndrome-constipation (IBS-C), for any number of days, at any dose, and at any time from the 1st day of the LMP up to and including the 12th week after the first day of the LMP. If the date of LMP is unclear, or if a first-trimester ultrasound has been done and the estimated date of conception is more than one week discrepant from the menstrual period calculation, the first-trimester ultrasound-derived date will be used to calculate a date for LMP and conception.
* Agree to the conditions and requirements of the study including the interview schedule, and release of medical records.

Cohort 2: Disease-Matched Comparison Cohort:

* Pregnant women.
* Diagnosed with CIC or IBS-C; frequency matched to the exposed group by disease indication, with the indication validated by medical records when possible.
* Agree to the conditions and requirements of the study including the interview schedule, and release of medical records.

Exclusion Criteria:

Cohort 1: Prucalopride-Exposed (MOTEGRITY, RESOTRAN) Cohort

* Women who have first contact with the project after prenatal diagnosis of any major structural defect.
* Women who have enrolled in the prucalopride cohort study with a previous pregnancy (women may only enroll once in the Prucalopride Pregnancy Cohort Study).
* Women who have used prucalopride for an indication other than CIC or IBS-C.
* Women who do not have exposure in the first trimester of pregnancy.
* Retrospective enrollment after the outcome of pregnancy is known (i.e. the pregnancy has ended prior to enrollment).
* Results of a diagnostic test are positive for a major structural defect prior to enrollment. However, women who have had any normal or abnormal prenatal screening or diagnostic test prior to enrollment are eligible as long as the test result does not indicate a major structural defect.

Cohort 2: Disease-Matched Comparison Cohort:

* Women who have first contact with the project after prenatal diagnosis of any major structural defect.
* Exposure to prucalopride (brand name or generic) anytime during the current pregnancy; may or may not have taken another medication for their disease in the current pregnancy.
* Women who have enrolled in the prucalopride cohort study with a previous pregnancy (women may only enroll once in the Prucalopride Pregnancy Cohort Study).
* Retrospective enrollment after the outcome of pregnancy is known (i.e. the pregnancy has ended prior to enrollment).
* Results of a diagnostic test are positive for a major structural defect prior to enrollment. However, women who have had any normal or abnormal prenatal screening or diagnostic test prior to enrollment are eligible as long as the test result does not indicate a major structural defect.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women from the United States (US) and Canada who have or have not been treated with prucalopride for CIC or IBS-C during their pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Major Structural Defects | Up to 1 year of age
  Major structural defects are defined and classified using the US Centers for Disease Control and Prevention (CDC) coding manual that is used for the Metropolitan Atlanta Congenital Defects Program (MACDP) classification of major structural defects. All major structural defects will be adjudicated by the co-investigator on this study.

SECONDARY OUTCOMES:
Number of Participants With Spontaneous Abortion/Miscarriage | 20 weeks post-last menstrual period (LMP)
  Spontaneous abortion/miscarriage is defined as non-deliberate fetal death that occurs prior to 20 weeks post-LMP.
Number of Participants With Stillbirth | From 20 weeks post-LMP to end of pregnancy
  Stillbirth is defined as non-deliberate fetal death anytime in gestation at or after 20 weeks post-LMP.
Number of Participants With Elective Termination/Abortion | At the end of pregnancy or through 9-month pregnancy period
  Elective termination/abortion is defined as deliberate termination of pregnancy through medication or surgical procedures. Elective abortions are classified for medical or social reasons.
Number of Participants With Premature Delivery | Through 9-month pregnancy period
  Premature delivery is defined as live birth prior to 37 weeks gestation as counted from LMP (or calculated from first-trimester ultrasound-derived due date if LMP uncertain or more than 1 week discrepant). Elective caesarian deliveries or inductions prior to 37 completed weeks will be considered separately.
Incidence of Small for Gestational Age | At birth
  Small for gestational age is defined as birth size (weight, length or head circumference) less than the 10th centile for sex and gestational age using standard pediatric CDC growth curves for full term or preterm infants.
Number of Participants With Postnatal Growth Deficiency | Up to 1 year of age
  Postnatal growth deficiency is defined as postnatal size (weight, length or head circumference) less than the 10th centile for sex and age using National Center for Health Statistics (NCHS) pediatric growth curves, and adjusted postnatal age for premature infants if the postnatal measurement is obtained at less than 1 year of age.
Screening for Neurodevelopmental Milestones | 1 year of age
  Screening for neurodevelopment performed using the Ages and Stages Questionnaire (ASQ). An abnormal score is defined in the scoring guidelines.
Incidence of Hospitalization in Live Born Children | Up to 1 year of age
  Hospitalizations is defined as any hospitalization of the infant within the first year of life after discharge following delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda; Study Director, Study Director — The Organization of Teratology Information Specialists
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as the data are subject to contractual (or consent) provisions that prohibit transfer to third parties.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/6091a2c8688ad8001f42fbc2